CLINICAL TRIAL: NCT06851793
Title: Investigation of Postural Parameters, Physical Functions, Balance and Quality of Life in Different Hip Pathologies
Brief Title: Investigating Postural Parameters in Different Hip Pathologies
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Esra ATEŞ NUMANOĞLU, Research Assistant - PT, PhD, Hacettepe University
Other Study IDs: SBA 24/191
Record Dates: First submitted 2024-10-28; First posted 2025-02-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hip Injuries and Disorders
Keywords: Hip Injuries and Disorders; Posture; Hip Functions; Physical Function; Pelvis
MeSH Terms: conditions — Hip Injuries; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with hip pathologies: Volunteers with hip pathology (hip osteoarthritis, hip impingement syndrome, hip labrum tear, hip dysplasia, hip avascular necrosis) who apply to the Orthopedic Rehabilitation Unit of the Faculty of Physical Therapy will be included in this group
- Healthy individuals: Healthy individuals between the ages of 18-65 who have been diagnosed with any of the following diagnoses: hip osteoarthritis, hip impingement syndrome, hip labrum tear, hip dysplasia, or hip avascular necrosis will be included in this group.

SUMMARY:
"It is known that pelvic parameters affect physical hip functions in hip pathologies. Depending on the type and severity of hip pathologies, posture, muscle strength, balance, and pain parameters may change, thereby impacting an individual's quality of life. This study aimed to examine the postural parameters, muscle strength, balance, quality of life, pain intensity, and pain localization of individuals with different hip pathologies, including hip osteoarthritis, hip impingement syndrome, hip labrum tear, hip dysplasia, and hip avascular necrosis."

DETAILED DESCRIPTION:
Volunteers with hip pathologies, such as hip osteoarthritis, hip impingement syndrome, hip labrum tear, hip dysplasia, and hip avascular necrosis, will be included in the study. Prior to the study, the responsible researcher will provide detailed face-to-face information regarding the study's content, the scales to be applied, the importance of these scales, and the evaluation processes. Individuals who agree to participate will sign an informed consent form before the evaluations begin. Demographic information will be recorded, and the dominant extremity for both the upper and lower extremities will be determined.

The measurements and evaluations will be conducted by the same researcher using a consistent evaluation method for all participants included in the study.

Volunteers with hip joint pathologies who apply to the Orthopedic Unit of Hacettepe University Faculty of Physical Therapy will be included in the study. During the initial interview, participants will be informed about the surveys and the parameters to be evaluated. The sample size was calculated using the G*Power 3.1 program, with an effect size of 0.74, an alpha error rate of 0.05, and a test power of 0.80. This included individuals with various hip pathologies (hip osteoarthritis, hip impingement syndrome, hip labrum tear, hip dysplasia, and hip avascular necrosis). The sample size for the study was determined to be 30 individuals with hip pathologies and 30 healthy individuals. To account for potential incomplete evaluations, a total of 66 participants, with an additional 10%, will be included.

Inclusion Criteria:

Diagnosed with one of the following: hip osteoarthritis, hip impingement syndrome, hip labrum tear, hip dysplasia, or hip avascular necrosis, experiencing mechanical impact on the hip joint, symptoms ongoing for at least 6 months, aged between 18 and 65 years

Exclusion Criteria:

Diagnosed with scoliosis by a physician, diagnosed with any developmental disorder (e.g., Scheuermann's/Calve disorder), diagnosed with a neurological and/or cognitive disease that may affect cognitive functions, diagnosed with inflammatory arthritis, underwent surgery on the spine or extremities, diagnosed with an infection (e.g., spinal tuberculosis) or tumor (e.g., multiple myeloma), epilepsy or use of antidepressants/attention-enhancing drugs.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with any of the following: hip osteoarthritis, hip impingement syndrome, hip labrum tear, hip dysplasia, hip avascular necrosis.
* Having mechanical impact on the hip joint
* Symptoms have been ongoing for at least 6 months
* Being between the ages of 18-65

Exclusion Criteria:

* Being diagnosed with scoliosis by a physician
* Being diagnosed with any developmental disorder (Scheuermann's/Calve Disorder etc.),
* Being diagnosed with a neurological and/or cognitive disease that may affect cognitive functions
* Being diagnosed with Inflammatory Arthritis
* Having undergone surgery on the spine and extremities,
* Getting diagnosed with Infection (Spinal Tuberculosis etc.), Tumor (Multiple Myeloma)
* Epilepsy, Antidepressant / Attention enhancing drug use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with different hip pathologies (hip osteoarthritis, hip impingement syndrome, hip labrum tear, hip dysplasia, hip avascular necrosis) who volunteered the participate the study
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2025-10-02 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Postural Parameter | Up to 4 weeks
  The postures of the participants will be evaluated using the 4-DIERS. In this method, white light lines (raster lines) are projected onto the participants' backs, and the curvature of these lines is used to create a 3D shape of the back. The patterns formed by these curved lines are detected by the camera. With the help of the software, the detected convex and concave regions allow for the immediate determination of anatomical landmarks and fixed points. A mathematical algorithm is used to reconstruct a three-dimensional model of the spine.

SECONDARY OUTCOMES:
Pain Threshold | Baseline
  The pain threshold evaluation with an algometer is a method used to assess an individual's sensitivity to pressure-induced pain. An algometer is a device that applies gradually increasing pressure to a specific point on the body until the subject perceives pain. This measurement is referred to as the pressure pain threshold (PPT) and is widely used in clinical and research settings to evaluate pain sensitivity in conditions such as musculoskeletal disorders, fibromyalgia, and chronic pain syndromes.
  Pain threshold values are typically recorded in kilograms per square centimeter (kg/cm²) or Newtons (N). The minimum pain threshold represents the lowest pressure at which pain is first perceived, while the maximum pain threshold indicates the highest tolerated pressure before withdrawal. The mean PPT is calculated based on multiple measurements at different anatomical sites to provide a more reliable assessment of an individual's pain sensitivity. Lower pain threshold values suggest high
Hip and Hip Related Pain | Baseline
  The Visual Analog Scale (VAS) is a widely used tool for assessing pain intensity and other subjective experiences, such as fatigue or discomfort. It consists of a 10-centimeter (100 mm) horizontal or vertical line, with endpoints representing "no pain" (0) on the left and "worst imaginable pain" (10 or 100) on the right. Patients mark a point on the line that best reflects their perceived pain intensity.
  The minimum VAS score is 0, indicating no pain, while the maximum score is 10 (or 100, depending on scaling), representing severe or unbearable pain. The mean VAS score is often calculated in studies to determine the average pain level within a group of patients. The scale is simple, quick to administer, and highly effective in capturing pain variations over time, making it a valuable tool in clinical practice and research for monitoring pain management and treatment outcomes.
Muscle Strength | Baseline
  The Lafayette Manual Muscle Dynamometer (Lafayette MMD) is a handheld device used to measure muscle strength in various muscle groups. It provides objective, quantifiable data on muscle force production, making it useful in rehabilitation, sports science, and clinical assessments of neuromuscular conditions. The device applies resistance to a specific muscle or muscle group while recording the maximum isometric force exerted by the patient.
  Muscle strength measurements with the Lafayette MMD are typically recorded in kilograms (kg) or Newtons (N). The minimum strength value represents the lowest recorded force, while the maximum strength value is the highest force exerted by the muscle during testing. The mean strength value is calculated to provide an overall assessment of muscle function. Higher values indicate greater muscle strength, whereas lower values may suggest muscle weakness or impairment, which is particularly relevant for patients undergoing rehabilitation or recovering
Hip Functions | Baseline
  The Harris Hip Score (HHS) is a clinician-based outcome measure used to assess the function, pain, and range of motion in patients undergoing hip surgery or suffering from hip disorders. The total score ranges from 0 to 100, with higher scores indicating better hip function. The HHS includes four main components: pain (44 points), function (47 points), absence of deformity (4 points), and range of motion (5 points). A score of 90-100 is considered excellent, 80-89 good, 70-79 fair, and below 70 poor.
Hip Functions | Baseline
  The Hip Outcome Score (HOS) is a patient-reported outcome measure designed primarily for younger, active individuals, especially those undergoing hip arthroscopy. It consists of two subscales: the Activities of Daily Living (ADL) subscale (17 items) and the Sports subscale (9 items). Each item is scored on a 0 to 4 scale, with 0 representing an inability to perform the activity and 4 indicating no difficulty. The total score is calculated as a percentage, with 100% representing the best possible function. The HOS is particularly useful for assessing hip function in active populations and tracking progress after surgical or non-surgical interventions.

OTHER OUTCOMES:
Balance | Up to 4 weeks
  The SENSAMOVE Balance Device is an advanced tool used for assessing and training balance, stability, and postural control. It utilizes sensor technology to provide real-time feedback on body movements, making it particularly useful in rehabilitation, sports training, and clinical assessments. The device measures shifts in weight distribution and postural sway, helping individuals improve their coordination and stability through targeted exercises.
  The balance performance scores from the SENSAMOVE device vary depending on the specific test protocols used. Typically, the device records minimum, maximum, and mean balance scores, which indicate the user's ability to maintain stability during different tasks. Higher scores generally reflect better balance control, whereas lower scores indicate greater postural instability.
Quality of Life Level | Baseline
  The SF-36 Quality of Life Scale (SF-36) is a widely used patient-reported outcome measure that assesses overall health and well-being across multiple dimensions. It consists of 36 items grouped into eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. These domains collectively provide a comprehensive assessment of an individual's physical and mental health status.
  Each domain of the SF-36 is scored on a 0 to 100 scale, with higher scores indicating better health and quality of life. In addition to the individual domain scores, the SF-36 can also generate two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS), which provide an overall view of physical and mental well-being. The mean scores vary across different populations and health conditions, but in general, a score closer to 1
Dominant extremity | Baseline
  The Waterloo Handedness and Footedness Questionnaire is a self-reported measure designed to assess an individual's preference for hand and foot usage in various tasks. It evaluates laterality by determining the degree to which a person favors one hand or foot over the other in everyday activities. The questionnaire consists of two separate sections, one for hand preference and another for foot preference, each containing multiple items that require individuals to indicate their preferred limb for specific tasks.
  The total scores for handedness and footedness range from -100 to +100, where -100 represents strong left-hand or left-foot preference, 0 indicates no preference (ambidextrous), and +100 signifies strong right-hand or right-foot preference. The mean scores vary based on population norms, but typically, a strong preference for either the left or right side results in scores closer to the respective extreme values. This questionnaire is commonly used in research on laterality,

CONTACTS AND LOCATIONS:
Overall Officials: Melike Naz GÜREL, MSc, Study Chair — Hacettepe University; Gürsoy COŞKUN, Prof, Study Chair — Hacettepe University; Esra ATEŞ NUMANOĞLU, PhD, Principal Investigator — Hacettepe University; Asude ARIK, PhD, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kechagias VA, Grivas TB, Papagelopoulos PJ, Kontogeorgakos VA, Vlasis K. Truncal Changes in Patients Suffering Severe Hip or Knee Osteoarthritis: A Surface Topography Study. Clin Orthop Surg. 2021 Jun;13(2):185-195. doi: 10.4055/cios20123. Epub 2021 Mar 16. PMID 34094009
- [Background] Jain M, Mohapatra A, Tripathy SK, Mohakud S, Das A, Sethy SS. Do Spinopelvic Parameters Relate with Secondary Hip Spine Syndrome in Secondary Hip Arthritis? Indian J Orthop. 2022 Sep 10;56(11):1937-1943. doi: 10.1007/s43465-022-00741-1. eCollection 2022 Nov. PMID 36310546
- [Background] Lanza MB, Arbuco B, Ryan AS, Shipper AG, Gray VL, Addison O. Systematic Review of the Importance of Hip Muscle Strength, Activation, and Structure in Balance and Mobility Tasks. Arch Phys Med Rehabil. 2022 Aug;103(8):1651-1662. doi: 10.1016/j.apmr.2021.12.008. Epub 2022 Jan 5. PMID 34998714
- [Background] Degenhardt BF, Starks Z, Bhatia S. Reliability of the DIERS Formetric 4D Spine Shape Parameters in Adults without Postural Deformities. Biomed Res Int. 2020 Feb 13;2020:1796247. doi: 10.1155/2020/1796247. eCollection 2020. PMID 32104678
- [Background] Mayne E, Memarzadeh A, Raut P, Arora A, Khanduja V. Measuring hip muscle strength in patients with femoroacetabular impingement and other hip pathologies: A systematic review. Bone Joint Res. 2017 Jan;6(1):66-72. doi: 10.1302/2046-3758.61.BJR-2016-0081. PMID 28108483
- [Background] Philippi MT, Kahn TL, Adeyemi TF, Maak TG, Aoki SK. Leg dominance as a risk factor for femoroacetabular impingement syndrome. J Hip Preserv Surg. 2020 Feb 13;7(1):22-26. doi: 10.1093/jhps/hnaa007. eCollection 2020 Jan. PMID 32382425
- [Background] Euasobhon P, Atisook R, Bumrungchatudom K, Zinboonyahgoon N, Saisavoey N, Jensen MP. Reliability and responsivity of pain intensity scales in individuals with chronic pain. Pain. 2022 Dec 1;163(12):e1184-e1191. doi: 10.1097/j.pain.0000000000002692. Epub 2022 May 18. PMID 35584261
- [Background] Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. J Strength Cond Res. 2009 Jan;23(1):312-4. doi: 10.1519/jsc.0b013e31818f051c. PMID 19130648
- [Background] Romero-Franco N, Jimenez-Reyes P, Montano-Munuera JA. Validity and reliability of a low-cost digital dynamometer for measuring isometric strength of lower limb. J Sports Sci. 2017 Nov;35(22):2179-2184. doi: 10.1080/02640414.2016.1260152. Epub 2016 Nov 24. PMID 27882825
- [Background] Polat G, Celik D, Cil H, Erdil M, Asik M. Evidence for reliability, validity and responsiveness of Turkish version of Hip Outcome Score. Acta Orthop Traumatol Turc. 2017 Jul;51(4):319-324. doi: 10.1016/j.aott.2017.05.001. Epub 2017 Jun 9. PMID 28602527
- [Background] Celik D, Can C, Aslan Y, Ceylan HH, Bilsel K, Ozdincler AR. Translation, cross-cultural adaptation, and validation of the Turkish version of the Harris Hip Score. Hip Int. 2014 Sep-Oct;24(5):473-9. doi: 10.5301/hipint.5000146. Epub 2014 Sep 10. PMID 25264204